CLINICAL TRIAL: NCT06359808
Title: A Study Based on the Microbiota-gut-brain Axis to Explore the Clinical Characteristics of Sleep Disorders in Patients With Ulcerative Colitis
Brief Title: Clinical Characteristics of Sleep Disorders in Patients With Ulcerative Colitis
Status: Recruiting | Type: Observational
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KY20232370
Record Dates: First submitted 2024-04-06; First posted 2024-04-11 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Colitis, Ulcerative; Sleep Quality; Gastrointestinal Microbiome; Autonomic Nervous System Imbalance
MeSH Terms: conditions — Colitis, Ulcerative; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Fecal, plasma and fixed tissue samples of some participants will be collected.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ulcerative colitis group: Ulcerative colitis patients aged 18-65 years will be recruited from The First Affiliated Hospital of the Air Forth Medical University from April 2024 to December 2024.
- Healthy subjects: Age-, gender-, and education level-matched healthy controls will be recruited from The First Affiliated Hospital of the Air Forth Medical University from April 2024 to December 2024.

SUMMARY:
Ulcerative colitis(UC) is one of the two main forms of inflammatory bowel disease(IBD), which seriously affects the quality of life of patients. Previous studies have demonstrated that more than 60% of IBD patients have sleep disorders, which is emerging as an important risk factor for disease recurrence and poor prognosis. However, the mechanisms by which sleep disorders regulates the occurrence and development of IBD remain undefined. This study aims to explore the clinical characteristics of ulcerative colitis patients with sleep disorders based on the microbiota-gut-brain axis, to analyze the effects of sleep disorders on autonomic nervous function, gut microbiota, and metabolites in UC patients.

DETAILED DESCRIPTION:
According to the inclusion and exclusion criteria, 152 UC patients of the First Affiliated Hospital of the Air Forth Medical University from April 2024 to December 2024 will be included. The PSQI scale was used to evaluate the sleep quality of the enrolled patients, and the overall incidence and severity of sleep disorders in UC patients will be evaluated. According to whether the PSQI score is higher than 5 points, the subjects will be divided into UC with sleep disorder group and the UC without sleep disorder group. By reviewing electronic medical records and questionnaire surveys, general clinical information of the subjects will be collected to analyze the risk factors of sleep disorders in UC patients. Mayo score and fecal calprotectin levels will be used to assess disease activity. The correlation between sleep disorders and disease activity in UC patients will be evaluated. Age-, gender-, and education level-matched healthy controls will be recruited from The First Affiliated Hospital of the Air Forth Medical University from April 2024 to December 2024. Heart rate variability will be measured to evaluate vagal nerve activity. Serum pancreatic peptide, norepinephrine, acetylcholine, and serotonin will be measured to evaluate serum neurotransmitter levels, and resting state functional magnetic resonance imaging will be used to evaluate the brain functional activity area of the subjects. Differences and correlations in autonomic nervous system function between UC with sleep disorder and UC without sleep disorder will be explored. 16s sequencing and metabolomics will be used to analyze changes in gut microbiota and metabolites. The correlation between gut microbiota and metabolites and sleep disorders in UC patients will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Ulcerative colitis was diagnosed according to the Consensus Opinions on the Diagnosis and Treatment of Inflammatory Bowel Disease (Beijing, 2018);
* Complete medical records and signed informed consent.

Exclusion Criteria:

* Previous mental illness or taking anti-anxiety and depression drugs;
* Patients with malignant tumors of digestive system or serious diseases of organs such as heart, lung, liver and kidney function damage or diseases of blood system;
* Drugs that affect heart rate or autonomic nervous function, such as glucocorticoids, beta-blockers, calcium channel blockers, etc. have been taken within the last 2 weeks;
* People who smoke, drink alcohol, drink tea, and drink coffee within 24 hours (all stimulants, which can easily lead to excitement and affect heart rate variability);
* Other diseases associated with autonomic nervous dysfunction (such as hyperthyroidism, hypertension, atrial premature beat, ventricular premature beat, pre-excitation syndrome, left bundle branch block, right bundle branch block, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ulcerative colitis patients aged 18-65 years were recruited from The First Affiliated Hospital of the Air Forth Medical University.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Pittsburgh Sleep Quality Index (PSQI) | At baseline
  PSQI is used to evaluate the sleep quality of the subjects in the last 1 month. There are 7 dimensions and 9 entries with a total score between 0 and 21, where a score higher than 5 indicates a sleep quality problem, 0 to 5 indicates good sleep quality, 6 to 10 indicates moderate sleep quality, 11 to 15 indicates poor sleep quality, and 16 to 21 indicates very poor sleep quality.
Disease activity | At baseline
  The modified Mayo score and calprotectin are used to assess the disease activity of ulcerative colitis patients.
Heart Rate Variability (HRV) | At baseline
  HRV reflects the continuous oscillations of the R-R intervals between normal heartbeats and is strongly correlated with actual vagal nerve activity. HRV thus provides a noninvasive and quantitative index of parasympathetic nervous system activity.
Functional Magnetic Resonance Imaging | At baseline
  Resting-state functional MRI (rs-fMRI) is a noninvasive imaging modality that is able to measure spontaneous low-frequency blood oxygen level-dependent signal fluctuations at rest to infer neuronal activity.
Neurotransmitter Agents | At baseline
  Serotonin, Pancreatic Polypeptide, Norepinephrine and Acetylcholine will be tested.
Gastrointestinal Microbiome | At baseline
  Fecal samples of some participants will be collected and prepared. DNA will be extracted from the stool samples, and the V3-V4 hypervariable region of bacterial 16S rRNA gene was sequenced.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | At baseline
  PHQ-9 is a widely used international universal depression screening scales. It consists of nine main entries, each with a score of 0 to 3 and a total score between 0 and 27.
Generalized Anxiety Disorder (GAD-7) | At baseline
  GAD-7 is a widely used anxiety screening scales. It includes 7 entries, each with a score of 0 to 3 and a total score between 0 and 21.
Inflammatory Bowel Diseases Questionnaire (IBDQ) | At baseline
  IBD-Q has been widely used to evaluate the quality of life of IBD patients, including 4 dimensions of bowel symptoms, systemic symptoms, emotional ability, and social ability, with a total of 32 items.18 Each item is divided into 7 levels, counting from 1 to 7, with 1 indicating the most severe degree and 7 indicating the least severe degree. The total score ranged from 32 to 224, and the higher the total score, the better the patient's quality of survival.

CONTACTS AND LOCATIONS:
Overall Officials: Kaichun Wu, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China